CLINICAL TRIAL: NCT00036153
Title: A Randomized, Double-Blind Study to Assess the Efficacy of Tacrolimus (Prograf®)+ Methotrexate Vs. Placebo + Methotrexate in the Treatment of Rheumatoid Arthritis in Patients With Partial Response to Methotrexate
Brief Title: Study to Assess Efficacy of Tacrolimus + Methotrexate Versus Placebo + Methotrexate in Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-0-103
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2011-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Tacrolimus, Prograf®, FK506
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus; Methotrexate

INTERVENTIONS:
Drug: Tacrolimus (Prograf®)
Drug: Methotrexate

SUMMARY:
The purpose of this study is to evaluate the efficacy of the combination of tacrolimus + methotrexate compared to methotrexate alone in the treatment of the signs and symptoms of rheumatoid arthritis over 6 months in patients with partial response to methotrexate.

DETAILED DESCRIPTION:
This is a Phase III, 6 month randomized, double-blind, placebo controlled multi-center study with a 6 month open-label extension. Patients will be randomized to the tacrolimus + methotrexate arm or the placebo + methotrexate arm in a ratio of 2:1. Patients who complete the 6-month double-blind phase will be eligible to enroll in the open-label phase of the study.

ELIGIBILITY:
Inclusion Criteria

* Willing to discontinue DMARDs, other than methotrexate
* Has a diagnosis of Rheumatoid Arthritis using American College of Rheumatology Criteria, of at least 6 months duration
* Have been receiving oral or parenteral methotrexate for at least 3 months

Exclusion Criteria

* Has received tacrolimus for any indication
* Has moderate or severe liver disease
* Has a known history of HIV infection
* Has serum creatinine outside the normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2002-03; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Radiant Research, Pharmaceutical Clinical Trials Division, Scottsdale, Arizona
  - Boling Clinical Trials, Rancho Cucamonga, California
  - San Diego Arthritis & Osteoporosis Medical Clinic, San Diego, California
  - Pacific Arthritis Center and Medical Group, Santa Maria, California
  - Arthritis Associates of CT, Danbury, Connecticut
  - Stamford Therapeutic Consortium, Stamford, Connecticut
  - Center of Rheumatology, Immunology & Arthritis, Fort Lauderdale, Florida
  - Arthritis Center, Palm Harbor, Florida
  - Sarasota Arthritis Center, Rheumatology Division, Sarasota, Florida
  - Arthritis & Rheumatology Associates of Palm Beach, West Palm Beach, Florida
  - Coeur d'Alene Arthritis Clinic, Coeur d'Alene, Idaho
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois Bone & Joint Institute, Morton Grove, Illinois
  - Rockford Clinical, Rockford, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Arthritis & Osteoporosis Center of Maryland, Frederick, Maryland
  - Phase III Clinical Research, Fall River, Massachusetts
  - Midwest Arthritis Center, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Arthritis Consultants, St Louis, Missouri
  - Arthritis Regional Research Center, Mercerville, New Jersey
  - New Jersey Physicians, LLC, Passaic, New Jersey
  - North Carolina Arthritis & Allergy Care Center, Raleigh, North Carolina
  - Radiant Research - Columbus, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - PRO Research, Eugene, Oregon
  - Oregon Health Sciences Center, Portland, Oregon
  - Portland Medical Associates, P.C., Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Center for Assessment & Research of Erie, Erie, Pennsylvania
  - Central Pennsylvania Clinical Research, Mechanicsburg, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Radiant Research - Dallas, Dallas, Texas
  - San Antonio Center for Clinical Research, San Antonio, Texas
  - Physicians Research Options, L.C., Sandy City, Utah
  - Metropolitan Clinical Research, Falls Church, Virginia
  - Lewis-Gale Clinic, Salem, Virginia
- Canada (2):
  - Doctor's Office, Hamilton, Ontario
  - The Arthritis Program Research Group, Inc., Newmarket, Ontario